CLINICAL TRIAL: NCT06604065
Title: Stimulation of Muscle Protein Synthesis With Essential Amino Acids in Parkinsons Disease
Brief Title: Essential Amino Acids and Parkinsons Disease
Acronym: EAAPD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EAAPD1
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMS2434 (amino acids) (Experimental): Product AMS2434. A single dose providing 10g of essential amino acids (EAAs).
  Study products will be in powder form and packaged in individual serving sizes and will be dissolved in 8 oz water for consumption.
  Interventions: Drug: AMS2434 (amino acids)
- Placebo (Placebo Comparator): Matched non-caloric placebo.
  Study products will be in powder form and packaged in individual serving sizes and will be dissolved in 8 oz water for consumption.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMS2434 (amino acids) — The proprietary composition includes leucine, valine, isoleucine, lysine, phenylalanine, threonine, tyrosine, histidine, and methionine. Small amounts of non-caloric flavorings are also included.
  Other Names: Amino Acids
  Arms: AMS2434 (amino acids)
Drug: Placebo — Matched non-caloric placebo. Study products will be in powder form and packaged in individual serving sizes and will be dissolved in 8 oz water for consumption.
  Arms: Placebo

SUMMARY:
Parkinson's disease is a neuromuscular disease that is relatively common in elderly that has many potentials symptoms, including a variety of physical features that together reduce quality of life. The Study Team have developed a nutritional supplement (AMS2434) based on essential amino acids that targets improving muscle health and brain neurotransmitter balance. This protocol will determine in individuals with PD the effect of AMS2434 on muscle protein synthesis, neurotransmitter production, and mood and cognition.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is characterized by the loss of dopaminergic neurons in the substantia nigra and is the second most common neurodegenerative disease in older individuals. PD may involve a variety of symptoms, but the predominant manifestation is impaired physical function, including muscle atrophy and weakness, bradykinesia, and reduced endurance. Older PD patients frequently present with, or develop, greater loss of muscle mass than expected from aging alone (sarcopenia). Sarcopenia results in inactivity, chronic inflammation, and neurodegeneration, all of which compound the loss of muscle function due to PD. L-DOPA/carbidopa is the most common drug therapy for PD and can mitigate some of the physical problems with PD, but progression of the disease usually ultimately results in severe reduction of quality of life.

The metabolic basis for loss of muscle mass with sarcopenia is anabolic resistance, defined as a diminished stimulation of muscle protein synthesis by dietary protein. Reduced muscle protein synthesis in response to dietary protein consumption not only contributes to the loss of muscle mass, but also to impaired single muscle fiber function, decreased mitochondrial biogenesis, and reduced neuromuscular junction stability, all of which contribute to impaired physical function. The consequences of anabolic resistance of muscle protein in PD is often compounded by the recommendation for reduced consumption of dietary protein due to the potential interference of absorbed dietary amino acids with the transport of L-DOPA from the intestine into the blood and from the blood into the brain.

We have developed an EAA-based nutritional supplement called AMS2434 designed to stimulate muscle protein synthesis in older individuals with PD and to promote dopamine production in the brain. AMS2434 is cleared rapidly from the blood after consumption, thereby minimally interfering with the transport of L-DOPA/carbidopa. In addition, AMS2434 contains tyrosine to enhance the brain production of dopamine. AMS2434 also decreases plasma tryptophan, which in turn reduces its degradation product kynurenine, which may be involved in the development of sarcopenia. We have previously shown that a 10g dose of EAAs maximally stimulates muscle protein synthesis in healthy elderly. In the current protocol we will determine if 10g of a mixture of a specifically designed mixture of EAAs (AMS2434) will robustly stimulate muscle protein synthesis in anabolic resistant individuals with Parkinson's disease. In addition, we will determine if AMS2434 stimulates brain dopamine synthesis from tyrosine.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Clinical diagnosis of idiopathic Parkinson Disease
* Hoehn and Yahr stage 2-3
* Stable medication regimen with L-DOPA/carbidopa for at least 4 weeks prior to study entry

Exclusion Criteria:

* Findings suggestive of atypical or secondary Parkinsonism, including cerebellar sign
* Use of anticoagulation drugs (including aspirin and Plavix) within one week of the protocol
* Allergy to lidocaine
* Supranuclear gaze palsy, apraxia, prominent autonomic failure, or other cortical signs
* Multiple strokes with stepwise progression of symptoms
* Neuroleptic treatment at time of study entry or time of onset of Parkinsonism
* Inability to walk without a cane or walker
* Deep brain stimulation
* Montreal Cognitive Assessment (MoCA) score <18
* Use of investigational drugs
* Early Alzheimer's disease
* Frontotemporal dementia of dementia with Lewy bodies
* Major depression treated with SSRIs
* Individuals with auditory or visual hallucinations
* Individuals taking drugs that cause Parkinsonism like symptoms such as antipsychotics, anti-emetics, prokinectic and anti-seizure medications

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 4 hours
  Mixed muscle protein synthesis expressed as the fractional synthetic rate.

SECONDARY OUTCOMES:
Whole body protein breakdown | 6 hours
  Amount of protein broken down per unit of time
Whole body protein synthesis | 6 hours
  Amount of protein gained per unit of time
Plasma concentrations of amino acids | 8 hours
  Measured via liquid chromatography mass spectrometry.
Plasma concentrations of kynurenine | 6 hours
  Measured via enzyme-linked immunosorbent assay
Plasma concentrations of homovanillic acid (HVA) | 6 hours
  Measured via enzyme-linked immunosorbent assay
Homovanillic acid (HVA) production from tyrosine | 6 hours
  Calculated from the isotopic enrichments of plasma HVA and tyrosine
D-KEFS color-word interference test | 6 hours
  Assessment of cognitive function
WAIS-IV symbol search | 6 hours
  Assessment of cognitive function
Trail making test | 6 hours
  Assessment of cognitive function
Profile of mood states (POMS) questionnaire | 6 hours
  Assessment of mood

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Wolfe, Ph.D., Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No